CLINICAL TRIAL: NCT03842956
Title: "Wound Closure (Allgower) Versus Secondary Open Wound Healing of the Pin Sites After Removal of the External Fixator: Study Protocol for a Prospective, Randomized Controlled Mono-center Trial"
Brief Title: Wound Closure (Allgower) Versus Secondary Open Wound Healing After Removal of the External Fixator
Acronym: Pinsides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Reto Babst, Head of Traumatology, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-01316
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Infection Rates Between Primary Wound-closure (Allgower) and Secondary Wound Healing After Removal of an External Fixator
Keywords: Fixator extern; Fixateur externe; External fixator; Wound healing; Fix-Ex; Pin Side; Trauma; Infection
MeSH Terms: conditions — Wounds and Injuries; Infections

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Blinded in the 6- and 52-weeks examination. So the doctor doesn't know which pin-side is treated by primary woundclosure (Allgower) or by secondary wound healing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary wound healing (Active Comparator): Primary woundclosure in Allgöwer suture technique
  Interventions: Procedure: Primary wound closure in Allgower Technique vs. secondary open wound healing of pin-sides after removal of the fixated-externe
- Secondary wound healing (No Intervention): no closure, open wound healing

INTERVENTIONS:
Procedure: Primary wound closure in Allgower Technique vs. secondary open wound healing of pin-sides after removal of the fixated-externe — We compare the outcome of primary wound closure (Allgower) and secondary open wound healing by comparing infection-rates, use of antibiotics, reoperation-rates, satisfaction of the patients and optical results using the Vancouver scar scale
  Arms: Primary wound healing

SUMMARY:
In this prospective randomized controlled single-center trial, based on a non-inferiority design, the outcome of the treatment of patients are analyzed, whereas in half of the cases the wounds are left open and the other ones are primary wound closed after local debridement after Fixator-Extern is removed. Although this topic embodies a daily business, there is no standard to be found in literature regarding the treatment of pin sites with closure by either primary or secondary intent.

DETAILED DESCRIPTION:
In the orthopedic department of the Kantonsspital Lucerne (LUKS) after removal of the external fixator, the pin sites at the tibia and the back of the foot are routinely treated with primary wound closure. An international survey carried out by the LUKS shows that in comparison to our standard treatment the majority of surgeons left the pin sites open during the healing process. In order to find a standardized method to treat pin sites we conduct a randomized controlled trial, in which half of the pin site wounds are left open and the other half are treated by primary wound closure after local debridement (Treatment of the first pin-side will be randomized, then alternated treatment of the consecutive pin-sides). All patients of the study participants are treated within a fixed pre- and postoperative protocol, which includes antibiotic prophylaxis with a single shot of Cefazolin 2g intravenously 30 minutes prior to surgery. The postoperative pin care includes daily inspection of the pin sites, cleaning the secondary healing wound with Ringerfundin © and disinfection with Betadine ©. Primary wound closures are dressed with dry gaze bandage. The following out-patient treatment is provided either by a Spitex support, the family doctor or by the patient himself, depending on the patients compliance. Regular follow-up consultations at 2, 6, 12, 24 and 52 weeks after surgery ensure an adequate surveillance of the healing process, whereas the examining doctor at the second and last consultation was kept in dark what therapy was chosen for pin sites of the patient. To objectify the clinical progress the pin sites are photo documented at the consultations at week 2 and 52.

ELIGIBILITY:
Inclusion Criteria:

* Completed 18th year of age
* Supply by external fixator
* Signed informed consent for study participation

Exclusion Criteria:

* Patients with immunodeficiency (HIV / hepatitis infection, leukemia, steroid therapy, autoimmune therapy)
* Patients who can not perform a follow-up treatment for structural reasons (tourists, not home canton) or other reasons
* Lack of knowledge of German
* Lack of consent to study participation
* invalid patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Post surgical pin side wound infections according to center of disease control (CDC) | up to 12 weeks after surgery

SECONDARY OUTCOMES:
Surgical wound revision of the pin sides, carried out antibiotic therapy in a wound infection | up to 52 weeks after surgery
Time to wound healing of the pin sides | up to 6 weeks after surgery
  Definition wound healing: complete epithelialization
Vancouver scar scale | up to 52 weeks after surgery
  ExercisingPigmentation 0-2, Vascularity 0-3, Pliability 0-5, Height 0-3, so that the score has got a total score reaching from 0 up to 13
subjective perception of the wounds | up to 52 weeks after surgery
  questionnaire on subjective preference of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tillmann F, Hoepelman RJ, Cagienard F, Link BC, Babst R, van de Wall BJM, Beeres FJP. Primary Closure or Secondary Wound Healing of Pin Sites After External Fixator Removal: A Single-Center Blinded Randomized Controlled Trial. J Bone Joint Surg Am. 2023 Feb 1;105(3):207-213. doi: 10.2106/JBJS.22.00234. Epub 2023 Jan 9. PMID 36622896
- [Derived] Roth F, Cagienard F, Link BC, Hodel S, Lehnick D, Babst R, Beeres FJP. Primary or secondary wound healing of the pin sites after removal of the external fixator: study protocol for a prospective, randomized controlled, monocenter trial. Trials. 2020 Feb 19;21(1):205. doi: 10.1186/s13063-020-4087-8. PMID 32075685